**Evaluation of SkillTalk for Autistic Young Adults** 

Statistical Analysis Plan

NCT06281171

11/19/2024

Data analysis was conducted by the statistician for the project, Dr. Elizabeth Baumler. The Co-Investigator cleaned and prepared the data for analysis.

First, descriptive analyses were used to describe the baseline characteristics of participating young adult populations, and to explore the data on all model variables at all follow up points for distributional assumptions and unanticipated patterns that might affect subsequent analyses.

Second, bivariate analyses were used to compare the baseline demographic and outcome characteristics of the intervention and control groups and to test for relationships between the outcome variable and potential covariates being measured. Variables associated with both the outcome and the study arms at p<0.15 in individual bivariate analyses were included in regression models. Regression models were used to assess intervention impact while adjusting for potential confounders. Third, multilevel regression (hierarchical or random coefficients regression) analyses were used to evaluate the studies primary hypotheses.